CLINICAL TRIAL: NCT00744575
Title: Assessment of a Specific Neurophysiological Brain Pattern in Patients Suffering From Chronic Back Pain
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: PhD Stefan Schmidt, University Hospital Freibung
Other Study IDs: 200/08
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2009-01

CONDITIONS: Back Pain
Keywords: back pain; eeg; chronic pain
MeSH Terms: conditions — Back Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Chronic Back Pain
- 2: Healthy Sex & Age Matched Controls

SUMMARY:
The purpose of this study is whether patients suffering from chronic back pain for more than one year will show a specific neurophysiological pattern in the EEG. This pattern is referred to as Thalamo-Cortical Dysrhythmia (TCD) and consists most likely of a self sustaining loop between the Cortex and Thalamus. This pattern has been found before in patients with very severe chronic pain. Specific lesions to the Thalamus result in a reduction of this pattern and decrease in pain. With this study the investigators will assess whether this pattern can be found in back pain patients of different types. Patients will be measured by EEG for the existence of TCD and will undergo detailed pain and psychological diagnostic.

DETAILED DESCRIPTION:
The neurophysiological processing of chronic pain is despite large efforts in the recent years still not well understood. However the so called cortical pain matrix describes cortical areas associated with the perception and processing of pain stimuli. Most studies identify second somatic area (SII), the insular regions, the anterior cingulated cortex (ACC) as well as the contralateral thalamus and the primary somatic area (SI) (Peyron, Laurent & Garcia-Larrea, 2000) as areas related to pain processing. In two recent publications by a Swiss research group (Sarnthein, Stern, Aufenberg, Rousson & Jeanmonod, 2006; Stern, Jeanmonod & Sarnthein, 2006) a dynamical EEG in the cortex pattern is described which is obvious related to chronic neurogenic pain. This pattern consists of an increase in EEG power and a shift of the dominant peak towards lower frequencies, mainly high theta (6-9 Hz). Source localization demonstrates that this overactivation mainly takes place in the areas of the cortical pain matrix. The authors argue that this pattern termed thalamocortical dysrhythmia is due to a thalamocortical loops initiated from the central lateral nucleus in the thalamus. This hypothesis is supported by the effects of a therapeutic lesion within the thalamus which led to (a) pain relief of 95% and to (b) the disappearance of the dysrhythmic pattern described above.

The investigators will set out to conduct a observational trial in order to determine pain related EEG characteristics in patients suffering from chonic back pain. Twenty four patients will be recruited for the study. A 64 channel high-resolution EEG and the following parameter will be recorded: Neuropathic Pain Questionnaire (Backonja and Krause 2003), EuroQol, BSI, Graded hronic pain scale(Klasen, Hallner, Schaub, Willburger & Hasenbring, 2004)pain (McGill Pain Questionnaire, VAS pain), and generic quality of life (Fragebogen zur Lebenszufriedenheit, Henrich & Herschbach, 1996).

An age and sex matched control group of healthy participants will be measured with the same method in order to compare whether the patients show a dysrhythmia pattern.

ELIGIBILITY:
Inclusion Criteria:

* Chronic back pain of at least one year duration
* Command of German language
* Age 18-70

Exclusion Criteria:

* Psychiatric disorders
* Immune suppression

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic back pain
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Difference in EEG signature and pain perception between groups | 25 months

SECONDARY OUTCOMES:
Quality of life, pain perception, neuropathic pain questionnaire, brief symptom inventory, life satisfaction | 25 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Schmidt, PhD, Principal Investigator — Universtiy Medical Center Freiburg
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Derived] Schmidt S, Gmeiner S, Schultz C, Lower M, Kuhn K, Naranjo JR, Brenneisen C, Hinterberger T. Mindfulness-based Stress Reduction (MBSR) as Treatment for Chronic Back Pain - an Observational Study with Assessment of Thalamocortical Dysrhythmia. Forsch Komplementmed. 2015;22(5):298-303. doi: 10.1159/000440687. Epub 2015 Oct 16. PMID 26565981
- [Derived] Schmidt S, Naranjo JR, Brenneisen C, Gundlach J, Schultz C, Kaube H, Hinterberger T, Jeanmonod D. Pain ratings, psychological functioning and quantitative EEG in a controlled study of chronic back pain patients. PLoS One. 2012;7(3):e31138. doi: 10.1371/journal.pone.0031138. Epub 2012 Mar 14. PMID 22431961